CLINICAL TRIAL: NCT03818620
Title: DermScan - Research in the Development of a New Type of Digital Dermatoscope for Skin Cancer
Brief Title: Research in the Development of a New Type of Digital Dermatoscope for Skin Cancer
Acronym: DermScan
Status: Active, not recruiting | Type: Observational
Sponsor: Barco NV (Industry)
Responsible Party: Sponsor
Other Study IDs: CI-PROT-0010; B322201732457 (Other: Belgian registration number); 80M0675 (Other: FAMHP Belgium)
Record Dates: First submitted 2019-01-23; First posted 2019-01-28 (Actual); Last update posted 2025-02-05 (Actual); Status verified 2025-02

CONDITIONS: Skin Cancer; Skin Diseases
MeSH Terms: conditions — Skin Neoplasms; Skin Diseases

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | Unapproved Device: Yes | US Export: No

INTERVENTIONS:
Device: Barco digital dermatoscope device images — Images of skin lesion taken with the Barco dermatoscope by site team member
Device: Reference standard dermatoscope device images — Images of skin lesion taken with a standard dermatoscope device (as part of standard care)

SUMMARY:
This is a multicenter prospective observational clinical investigation with a medical device. The purpose of this study is to develop and validate of a new type of digital dermatoscope with automatic decision support algorithms. By means of this study a better insight can be gained of the current performance and workflow in clinical dermatoscopy. This knowledge will be used to further improve the developed technology.

ELIGIBILITY:
Inclusion Criteria:

* The patient has a lesion that is accessible to the Barco Digital Dermatoscope
* Patient gives informed consent
* Men or women of any ethnic group aged ≥ 18 years

Exclusion Criteria:

* Men or women of any ethnic group aged < 18 years
* Patients not willing or able to read, understand and sign the study-specific informed consent form

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients will be considered for enrollment in the study when they have a lesion that is accessible to the Barco Digital Dermatoscope, are able to give informed consent and are over 18 years old.
Sampling Method: Probability Sample
Enrollment: 3000 (Estimated)
Dates: Start 2017-06-07 (Actual); Primary Completion 2025-04-30 (Estimated); Study Completion 2025-04-30 (Estimated)

PRIMARY OUTCOMES:
Development of anonymized database with over 3000 (potential) skin cancer cases for use in AI | 3.5 years
  Database of multispectral images of potential skin cancer lesions acquired with the Barco device together with clinical information (e.g. age, gender, history of skin cancer, histopathology diagnosis) and matched standard images using medical photography

SECONDARY OUTCOMES:
Comparison of new device to standard dermoscopy | 2 years
  Compare clinical performance and workflow efficiency of the Barco device to current standard of care (standard dermoscopy)

CONTACTS AND LOCATIONS:
Overall Officials: Marjan Garmyn, Prof. Dr., Principal Investigator — UZ / KU Leuven; Lieve Brochez, Prof. Dr., Principal Investigator — UZ Gent
Locations (2):
- Belgium (2):
  - UZ Gent, Ghent
  - UZ / KU Leuven, Leuven

IPD SHARING:
Plan to Share IPD: No